CLINICAL TRIAL: NCT05078385
Title: A Pilot Safety Study of Mesenchymal Stem Cell Derived Extracellular Vesicles for the Treatment of Burn Wounds.
Brief Title: Safety of Extracellular Vesicles for Burn Wounds
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aegle Therapeutics (Industry)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGLE-102-102
Record Dates: First submitted 2021-10-12; First posted 2021-10-14 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AGLE-102 (Experimental): AGLE-102, bone marrow mesenchymal stem cell derived extracellular vesicles (EVs)
  Interventions: Drug: AGLE-102

INTERVENTIONS:
Drug: AGLE-102 — AGLE-102, bone marrow mesenchymal stem cell derived extracellular vesicles (EVs)

SUMMARY:
Treatment of patients with deep second degree burns of the skin with extracellular vesicles (EV) isolated from bone marrow derived mesenchymal stem cells.

DETAILED DESCRIPTION:
This study is designed to examine the safety and efficacy, in 10 patients of administration of allogeneic MSC EV to deep second degree burn wounds. The dose level delivered will be approximately 1 X 107 EV particles for each cm2 treated area. Wounds eligible for treatment will not exceed 600 cm2 per wound or collection of wounds in a defined anatomical area (e.g., arm, leg, chest) treated. Patients with 20% or greater TBSA in total (3700 cm2 in a 70 kg, 175 cm subject) will be ineligible to participate in the study. The first treatment will be administered within 48 hours of the burn injury. Two additional administrations of EV will be given approximately one week (day 5-7 post-injury) and two weeks after the first treatment (unless the wound is fully closed, in which case the patient will continue to be monitored at weekly intervals through 5 weeks, then at 8, 12, 26, and 54 weeks). Safety will be assessed by collection of adverse event data. The potential for wound healing efficacy will be evaluated by recording the percent of burns re-epithelialized within 8 weeks as well as the time to complete closure. Wound closure will be defined as complete re-epithelialization that is not subject to re-injury during dressing changes or as a result of normal daily activities (e.g., wearing clothing, eating, sleeping). The potential for tissue regeneration and restoration of pigmentation, hair growth and skin texture will be evaluated by scoring healing and scar formation using POSAS. Assessment of the potential for prevention of conversion will be done using LDI. Deep second degree wounds presenting at screening that are assessed to be deeper by LDI at the 5-7 day reading than at the initial evaluation in the first 72 hours will be considered to have undergone conversion. Exploratory endpoints will include monitoring for the presence of an immunologic response in recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Eighteen years of age or older with deep second degree thermal burn wounds
2. Index burn injury within the prior 72 hours
3. Subjects must understand and be willing and able to give written informed consent
4. Subjects must agree to have blood draws performed per protocol
5. Subjects must be accessible for wound treatment and assessment visits
6. Males and females must agree to use an acceptable method of contraception. Exceptions will be females of non-childbearing age and monogamous males who are partners of females of non-childbearing age. Acceptable methods of birth control include; history of sterilization, oral contraceptives, depo-progesterone injections, a barrier contraceptive such as a condom with or without spermicide cream or gel, diaphragms or cervical cap with or without spermicide cream or gel, or an intrauterine device (IUD).
7. Maximum index wound size at screening limited to single or multiple wounds (in a defined anatomical area) cumulatively ≤ 600 cm2. Minimum wound size at screening: 30 cm2. Other wounds may be present that are treated separately from this protocol subject to the maximum TBSA exclusion criteria listed below.

Exclusion Criteria:

1. Solely first degree or solely third degree burns
2. Cumulative burn area ≥ 20% TBSA (20% TBSA corresponds to 3700 cm2 in a 70 kg, 175 cm subject)
3. Burns that occur over a previous scar
4. Chemical, radiation, or electrical burns
5. Subjects with superficial second degree burn who are expected to heal within 2 weeks with standard therapy
6. Evidence of active infection at the wound site
7. Evidence of significant wound healing prior to treatment
8. Burn wounds requiring surgery (other than debridement), or skin grafting
9. Wound exclusively located in the area of fingers, toes, face, or perineum
10. Wound that extends > 50% across one or more joints
11. Have any requirement for the use of systemic steroids or immunosuppressive medications
12. Subjects allergic to human albumin, streptomycin, or penicillin
13. Be a pregnant female or nursing mother
14. Subjects who are known or found to be HIV positive
15. History of alcohol or substance abuse requiring treatment within the past 12 months.
16. Severe medical conditions

    1. Malignancy (other than non-melanoma skin cancer) not in remission or in remission less than 5 years
    2. Life expectancy less than two years
    3. Severe cardiopulmonary disease restricting ambulation to the clinical facility
17. WBC <3 or > 20 x109/L, Hgb < 9g/dL, platelet count 100x109/L or less, serum creatinine > 1.5 times the upper normal limit, AST or ALT > 2.4 times upper normal limit
18. Known history of coagulopathy
19. Subjects who have a reasonable likelihood of being a recipient of tissue or organ transplantation
20. History of poor compliance, unreliability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Examine the safety of applying up to three applications of EVs to deep 2nd degree burn wounds up to 600 cm2 | 1 year
  Examine the safety of applying up to three applications of EVs to deep 2nd degree burn wounds up to 600 cm2 by evaluating the number of participants with treatment-related adverse events as assessed cy CTCAE v4.0

SECONDARY OUTCOMES:
Determine if administration of EVs can promote wound healing by serial wound measurements | 8 weeks
  Determine if administration of EVs can promote wound healing by serial wound measurements; tissue regeneration as evidenced by restoration of pigmentation and hair growth by serial photography; and skin texture assessment the Patient and Observer Scar Assessment Scale (scale of 1 to 10, where 10 is a worse outcome).
Laser Doppler will assess differences in dermal perfusion rates between control (unburned) and treated burn tissues. | 1 year
  Laser Doppler will assess differences in dermal perfusion rates between control (unburned) and treated burn tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Schulman, MD, Principal Investigator — Ryder Trauma Center
Locations (2):
- United States (2):
  - Ryder Trauma Center, Miami, Florida
  - North Carolina Jaycee Burn Center, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No